CLINICAL TRIAL: NCT06438614
Title: A Phase II Single Center Study Of Naxitamab , Granulocyte Macrophage Colony Stimulating Factor (GM CSF and Ifosfamide Carboplatin Etoposide) For Patients With Relapsed Refractory , Soft Tissue or Anti GD2 Immunotherapy Refractory Neuroblastoma
Brief Title: A Study Of Naxitamab , Granulocyte Macrophage Colony Stimulating Factor For Patients With Relapsed /Refractory , Soft Tissue or Anti GD2 Immunotherapy Refractory Neuroblastoma
Acronym: NICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSJD HR NB.2 2019
Record Dates: First submitted 2024-03-21; First posted 2024-06-03 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-03

CONDITIONS: Refractory Neuroblastoma; Soft Tissue Cancer
MeSH Terms: conditions — Neuroblastoma; Sarcoma | interventions — naxitamab

STUDY DESIGN:
Intervention Model Description: Subjects will receive 2 cycles of HITS. Each cycle of HITS (4 doses of hu3F8, 5 doses of irinotecan and temozolomide and 5 doses of GM-CSF). Patients with CR after 2 or 4 cycles of HITS will receive 5 cycles of Naxitamab + GM-CSF cycles. Patients that do not have an objective response (CR/PR) will receive NICE within 3 weeks from last dose. Each cycle of NICE consists of 4 doses of hu3F8, 5 doses of GM-CSF, 1 dose of carboplatin, and 3 doses each of ifosfamide and etoposide. Patients with less than CR response (PR/SD) will receive 2 more cycles of NICE and evaluated after 4th cycle. Patients with no objective response at these timepoints will be removed from the study. Patients with CR will receive 5 cycles of Naxitamab consolidation cycles consisting of GM-CSF250mcg/m2/day SC administered from day -4 to day 0 and GM-CSF500mcg/m2/day SC administered from day 1 to day 5. Three doses of hu3F83 mg/kg IVwill be administrated, specifically on days 1, 3 and 5.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm 1 (Experimental): Treatment involves 2 cycles of HITS: hu3F8, irinotecan, temozolomide, and GM-CSF. Irinotecan and temozolomide are given for 5 days, and hu3F8 and GM-CSF on specific days.
  Following this, 5 cycles of Naxitamab + GM-CSF are administered. Patients without a response receive NICE: hu3F8, GM-CSF, carboplatin, ifosfamide, and etoposide for 4 cycles.
  Patients with a complete response (CR) move to Naxitamab consolidation (5 cycles). This involves GM-CSF before and after, and hu3F8 on days 1, 3, and 5.
  Those with less than CR undergo 2 more NICE cycles, evaluated after the 4th. Lack of response leads to removal from the study.
  Interventions: Drug: HITS; Drug: Naxitamab + GM-CSF cycles; Drug: NICE

INTERVENTIONS:
Drug: HITS — Four doses of hu3F8, five doses each of irinotecan and temozolomide and five doses of GM-CSF. Irinotecan 50mg/m2/day IV will be administered from day 1-5concurrently with temozolomide 150mg/m2/day orally. Hu3F8 2.25mg/kg IV will be administered on days 2, 4, 9and11. GM-CSF 250mcg/m2/day SC will be administered on days 7-11
Drug: Naxitamab + GM-CSF cycles — Patients that achieve CR after 2 or 4 cycles of HITS will move on to 5 cycles of Naxitamab + GM-CSF cycles.
Drug: NICE — Patients that do not have an objective response (CR/PR) will receive NICE within 3 weeks from last dose. Each cycle of NICE consists of four doses of hu3F8, five doses of GM-CSF, one dose of carboplatin, and 3 doses each of ifosfamide and etoposide (table 2). Hu3F8 2.25mg/kg IV will be administered on days 2, 4, 9and 11. GM-CSF 250mcg/m2/day SC will be administered on days 7-11. Ifosfamide 1.5 gr/m2/day IV will be administered from day 1-3 concurrently with etoposide 100 mg/m2/day IV. Carboplatin 400 mg/m2/day IV will be administered on day 1

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of naxitamab, granulocyte macrophage Colony Stimulating Factor (GM CSF) and Isofosfamide/Carboplatin/Etoposide (NICE) for Patients With Relapsed /Refractory, soft tissue or anti GD2 immunotherapy refractory Neuroblastoma

DETAILED DESCRIPTION:
The anti-GD2 monoclonal antibody Naxitamab (also known as hu3F8) in combination with macrophage colony-stimulating factor (GM-CSF) is currently under pivotal phase 3 investigation for the treatment of High-Risk Neuroblastoma Patients with Primary or Secondary Refractory Osteomedullary Disease.

A subset of patients with high-risk, resistant disease, i.e., relapsed or refractory Neuroblastoma with soft tissue involvement as measured by 123I-Meta-iodobenzylguanidine (MIBG), 18F-FDG avid or measurable computed tomography (CT)/ magnetic resonance imaging (MRI) tumors outside of the bone marrow, or disease refractory to Naxitamab in combination with GM-CSF has shown significant response rates to a chemoimmunotherapy combination of Naxitamab, GM-CSF, irinotecan and temozolomide (HITS- Hu3F8, irinotecan, temozolomide and sargramostim) (NCT03189706). Treatment is administered on an outpatient basis and toxicities include those expected from I/T (myelosuppression and diarrhea) as well as pain and hypertension expected with Naxitamab. No other greater than grade 2 related toxicities occurred in this study (n=46). Early responses, assessed after 2 cycles, were documented in 18 (39%) patients and here complete (n = 9), partial (n = 8), and mixed (n = 1) and 13 patients had stable disease. Responses were achieved in refractory (3/7;43%) and progressive disease (15/39;38%) subgroups, in patients who had previously received I/T (12/34;35%) and/or anti-GD2 MoAb (14/36;39%), and in soft tissue (6/22; 27%) MIBG-avid skeletal sites (20/36;56%) and on bone marrow histology (9/12;75%). While encouraging, new strategies are warranted to further treat resistant disease.

A high-dose combination of ifosfamide, carboplatin, and etoposide (ICE) has activity against Neuroblastoma without cross-resistance to widely used chemotherapy regimens.

Through compassionate use, 4 patients with progression of disease or refractory disease after HITS therapy, have been further treated with two cycles of a combination of naxitamab, Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) and ifosfamide/Carboplatin/Etoposide (NICE). The first patient showed a complete response.

Toxicity included G2 prolonged aplasia and G3 hypertension, both expected from the chemotherapy agents and hu3F8. One patient progressed after the 2 cycles and the other 2 showed stable disease, according to the revised (2017) International Neuroblastoma Response Criteria (INRC).

In this formal trial, the investigators will investigate whether the combination of Naxitamab and GM-CSF with ifosfamide/Carboplatin/Etoposide (ICE) has a synergistic treatment effect in relapsed or refractory disease. The safety and efficacy of NICE (Naxitamab, Ifosfamide/Carboplatin/Etoposide) in patients that have not achieved complete remission with HITS chemo-immunotherapy will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of neuroblastoma (NB) as defined per INRC as

   1. histopathology of tumor biopsy, or
   2. BM aspirate or biopsy indicative of NB by histology plus high blood or urine catecholamine metabolite levels or MYCN amplification, or
   3. Fluorodeoxyglucose (FDG), MIBG avid lesion(s)
2. High-risk NB as defined as any of the following:

   1. Stage 4 with MYCN amplification
   2. Stage 4 without MYC amplification >1.5 y of age
   3. Stage 3 with MYCN amplification
3. Relapsed/refractory Neuroblastoma with

   1. Evidence of soft tissue disease or
   2. Progessive disease/incomplete response/relapsed to previous treatment with Naxitamab plus GM-CSF
4. Prior treatment with murine and hu3F8 is allowed
5. Prior treatment with irinotecan or temozolomide or ICE is permitted
6. Evaluable (microscopic marrow metastasis, elevated tumor markers, positive MIBG or PET scans) or measurable (CT, MRI) disease documented after completion of prior systemic therapy
7. Age ≥18 months
8. Acceptable hematological status defined as:

   1. Hemoglobin ≥8 g/dL (5.0 mmol/L)
   2. White blood cell count ≥1000/μL
   3. Absolute Neutrophil Count (ANC) ≥500/μL
   4. Platelet count ≥50,000/μL
9. Acceptable liver function defined as:

   1. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5 times Upper Limit of Normal (ULN)
   2. Bilirubin ≤1.5 x ULN
10. Acceptable kidney function defined as:

    a. estimated Glomerular Filtration Rate (eGFR) >60 mL/min/1.73 m2 calculated by the 2009 revised Bedside Schwartz Equation
11. Written informed consent from legal guardian(s) and/or patient in accordance with local regulations. Children must provide assent as required by local regulations (≥ 12 years old).

Exclusion Criteria:

1. Existing major organ dysfunction > grade 2, with the exception of hearing loss and hematologic toxicity (defined as suppression of all subtypes of WBCs, RBCs, and platelets).
2. Active life-threatening infection.
3. Pregnant women or women who are breast-feeding.
4. Inability to comply with protocol requirements, including genetic studies.
5. History of allergy to GM-CSF ≥ G4 (Common Terminology Criteria for Adverse Events- CTCAE) or does not respond to treatment.
6. Absolute Neutrophil Count (ANC) < 500/uL .
7. Platelet count <50,000/uL.
8. Patients with relapsed/refractory Neuroblastoma with solely bone marrow/bone involvement. Only patients with B/BM compartiment disease who show progressive disease/incomplete response/relapsed to previous treatment with Naxitamab plus GM-CSF may be eligible (inclusion critèrium #3).

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | 14 months after ICF signature
  The safety and tolerability of the treatment will be determined by means of type, incidence, severity, timing, seriousness, and relatedness of reported AEs, physical examinations, and laboratory tests. Toxicity will be graded and tabulated by the NCI CTCA E v 5 .0
Best Overall Response (at the end of HITS treatment) | From first day of treatment with HITS until completion of HITS (39 days).
  Best Overall Response is defined as the best response recorded from the start of the study treatment
Best Overall Response of Complete Response (CR) (at the end of HITS treatment) | From first day of treatment with HITS until completion of HITS(39 days).
  The number and proportion of patients with CR as Best Overall Response at the end of HITS treatment
Objective Response Rate (at the end of HITS treatment) | From first day of treatment with HITS until completion of HITS (39 days).
  Objective Response Rate is defined as the proportion of patients with Best Overall Response of CR (complete response) or PR (partial response).
Clinical Benefit Rate (at the end of HITS treatment) | From first day of treatment with HITS until completion of HITS (39 days).
  Clinical Benefit Rate is defined as the proportion of patients with Best Overall Response of CR (complete response) or PR (partial response) or SD (stable disease) ≥ 24 w
Best Overall Response (at the end of NICE treatment) | From first day of treatment with NICE until completion of NICE (39 days).
  Best Overall Response is defined as the best response recorded from the start of the study treatment
Best Overall Response of Complete Response (CR) (at the end of NICE treatment) | From first day of treatment with NICE until completion of NICE (39 days).
  The number and proportion of patients with CR as Best Overall Response at the end of NICE treatment
Objective Response Rate (at the end of NICE treatment) | From first day of treatment with NICE until completion of NICE (39 days).
  Objective Response Rate is defined as the proportion of patients with Best Overall Response of CR (complete response) or PR (partial response).
Clinical Benefit Rate (at the end of NICE treatment) | From first day of treatment with NICE until completion of NICE (39 days).
  Clinical Benefit Rate is defined as the proportion of patients with Best Overall Response of CR (complete response) or PR (partial response) or SD (stable disease) ≥ 24 w

SECONDARY OUTCOMES:
To evaluate serum cytokines in patients receiving NICE | From first day of treatment with NICE, until day 11 post administration.
To measure MRD after HITS | From first day of treatment with HITS until completion of HITS (39 days).
  Minimal residual disease for NB will be evaluated using the Revised International NB Response Criteria (JCO August 1, 2017)
To measure MRD after NICE | From first day of treatment with NICE until completion of NICE (39 days).
  Minimal residual disease for NB will be evaluated using the Revised International NB Response Criteria (JCO August 1, 2017)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No